CLINICAL TRIAL: NCT07348159
Title: Efficacy of Nalbuphine in Attenuation of Hemodynamic Response to Laryngoscopy and Orotracheal Intubation: A Randomized Controlled Trial
Brief Title: Effect of Nalbuphine on Hemodynamic Response During Laryngoscopy and Intubation
Acronym: NAL-HRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Waseem Ullah (Other Government)
Collaborators: Hayatabad Medical Complex (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Waseem Ullah, Assistant Professor, Lady Reading Hospital, Pakistan
Organization: Lady Reading Hospital, Pakistan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMC-GAD-F 2231
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hemodynamic Response to Laryngoscopy and Orotracheal Intubation
Keywords: Nalbuphine; Laryngoscopy; Orotracheal Intubation; Mean Arterial Pressure; Hemodynamic Response; General Anesthesia; Opioid Premedication
MeSH Terms: interventions — Nalbuphine

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups to receive either intravenous nalbuphine or placebo prior to induction of general anesthesia.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation. Study drugs were prepared by personnel not involved in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Normal Saline) (Placebo Comparator): Participants in this arm received intravenous normal saline in a volume equivalent to the intervention drug. The placebo was administered five minutes before induction of general anesthesia, followed by standardized induction with propofol and atracurium, laryngoscopy, and orotracheal intubation.
  Interventions: Drug: Normal saline IV
- Nalbuphine 0.2 mg/kg (Experimental): Participants in this arm received intravenous nalbuphine at a dose of 0.2 mg/kg administered five minutes before induction of general anesthesia. Induction was standardized using propofol and atracurium, followed by laryngoscopy and orotracheal intubation.
  Interventions: Drug: Nalbuphine 0.2 mg/kg

INTERVENTIONS:
Drug: Normal saline IV — Intravenous administration of normal saline in a volume equivalent to the nalbuphine dose, 5 minutes prior to induction of general anesthesia for elective surgery. This serves as a placebo control to compare the effect of nalbuphine on attenuation of the hemodynamic response (mean arterial pressure and heart rate) during laryngoscopy and orotracheal intubation. Standard monitoring is applied during the procedure. Any adverse events are recorded similarly to the experimental group.
  Arms: Placebo (Normal Saline)
Drug: Nalbuphine 0.2 mg/kg — Intravenous nalbuphine at a dose of 0.2 mg/kg administered 5 minutes prior to induction of general anesthesia for elective surgery. The purpose of administration is to attenuate the hemodynamic response, specifically mean arterial pressure and heart rate changes, associated with laryngoscopy and orotracheal intubation. Standard monitoring is applied during the procedure, including continuous ECG, non-invasive blood pressure, pulse oximetry, and capnography. Any adverse events such as mild bradycardia or nausea are recorded.
  Arms: Nalbuphine 0.2 mg/kg

SUMMARY:
Laryngoscopy and placement of a breathing tube during general anesthesia can cause temporary increases in blood pressure and heart rate. These changes may be harmful in some patients. Nalbuphine is an opioid pain medicine that may reduce these cardiovascular responses.

This study evaluated whether intravenous nalbuphine, given before anesthesia induction, reduces changes in mean arterial blood pressure during laryngoscopy and orotracheal intubation compared with placebo (normal saline).

Adult patients undergoing elective surgery under general anesthesia were randomly assigned to receive either nalbuphine or placebo before anesthesia. Blood pressure was measured before drug administration, during intubation, and for several minutes afterward. The results of this study may help guide safe medication use to maintain blood pressure stability during airway management.

DETAILED DESCRIPTION:
Laryngoscopy and orotracheal intubation are essential components of general anesthesia but are associated with a sympathoadrenal stress response caused by stimulation of the laryngeal and pharyngeal structures. This response may result in transient hypertension and tachycardia due to catecholamine release. Although often well tolerated in healthy individuals, these hemodynamic changes can be undesirable and potentially harmful, particularly in patients with limited cardiovascular reserve.

Opioids have been widely used to attenuate the hemodynamic response to airway manipulation. Nalbuphine is a synthetic opioid with kappa receptor agonist and mu receptor antagonist properties. It provides analgesia with a ceiling effect on respiratory depression and has a lower risk of certain opioid-related adverse effects compared with pure mu agonists. Despite these potential advantages, data regarding the effectiveness of nalbuphine in attenuating intubation-related hemodynamic responses remain limited.

This prospective, randomized, controlled trial was conducted at Hayatabad Medical Complex, Peshawar, Pakistan, between March 2024 and December 2024. Adult patients aged 18 to 60 years with American Society of Anesthesiologists (ASA) physical status I, scheduled for elective surgery under general anesthesia requiring orotracheal intubation, were enrolled. Patients with anticipated difficult airways, cardiovascular disease, hypertension, hepatic or renal disease, pregnancy, opioid allergy, or use of interacting medications were excluded.

Eligible participants were randomly allocated into two groups. The intervention group received intravenous nalbuphine at a dose of 0.2 mg/kg, while the control group received an equivalent volume of normal saline. The study drug was administered five minutes before induction of anesthesia. Anesthesia induction was standardized using propofol and atracurium, followed by Macintosh laryngoscopy and orotracheal intubation performed by experienced anesthetists.

Hemodynamic parameters were recorded at baseline, three minutes after administration of the study drug, immediately after intubation, and at one-minute intervals for five minutes following intubation. The primary outcome measure was mean arterial pressure after laryngoscopy and intubation. Adverse events, including bradycardia, hypotension, nausea, respiratory depression, and other complications, were monitored intraoperatively.

The purpose of this study was to determine whether nalbuphine premedication provides better attenuation of the hemodynamic response to laryngoscopy and intubation compared with placebo in healthy adult patients undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for elective surgery under general anesthesia requiring laryngoscopy and orotracheal intubation.

American Society of Anesthesiologists (ASA) physical status I or II. Age between 18 and 60 years. Both male and female patients. Patients who provide written informed consent.

Exclusion Criteria:

Known hypersensitivity to nalbuphine or any opioids. History of cardiovascular disease, including uncontrolled hypertension, arrhythmias, or ischemic heart disease.

Patients with respiratory disorders such as asthma, chronic obstructive pulmonary disease, or significant respiratory compromise.

Patients with renal or hepatic impairment. Pregnant or lactating women. Patients on medications affecting hemodynamic response (e.g., beta-blockers, calcium channel blockers).

Emergency surgeries. Patients with anticipated difficult airway (Mallampati class III or IV).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Mean Arterial Pressure (MAP) change following laryngoscopy and orotracheal intubation | Immediately after intubation and at 1-minute intervals for 5 minutes post-intubation
  MAP will be measured at baseline (before drug administration), 3 minutes after administration of nalbuphine or placebo, immediately after intubation, and at 1-minute intervals for the subsequent 5 minutes. The primary outcome is the difference in MAP between the nalbuphine group and the saline control group, reflecting the efficacy of nalbuphine in attenuating the hemodynamic response to laryngoscopy and intubation.

SECONDARY OUTCOMES:
Heart Rate (HR) change | Immediately after intubation and at 1-minute intervals for 5 minutes post-intubation
  HR will be recorded alongside MAP at the same time points. The difference between groups will indicate the effect of nalbuphine on tachycardia associated with airway manipulation.
Incidence of adverse events | Intraoperative and immediate postoperative period
  Adverse events such as mild bradycardia (HR 50-55 bpm), hypotension (MAP <60 mmHg), transient hypertension (MAP >110 mmHg), nausea, respiratory depression, and allergic reactions will be recorded. The frequency and severity of these events will be compared between nalbuphine and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hayatabad Medical Complex, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, study protocol, and statistical analysis plan will be made available upon reasonable request to researchers after publication of the study results, for a period of 5 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will be available starting 6 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Access will be granted to researchers with a scientifically sound proposal. Data will be provided after approval of the request and signing of a data use agreement. Researchers will have access to de-identified participant data, study protocol, SAP, and ICF.